CLINICAL TRIAL: NCT05119140
Title: Administration of Hydroxychloroquine (Plaquenil) to African Americans and Hispanics for the Treatment of Mild to Severe Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Judy Cho, Dean of Translational Genetics, Director, The Charles Bronfman Institute for Personalized Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 20-0187
Record Dates: First submitted 2021-10-20; First posted 2021-11-12 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis (Disorder)
Keywords: Ulcerative Colitis; Plaquenil; Hydroxychloroquine; CTLA-4; Inflammatory Bowel Disease; Non European Ancestry
MeSH Terms: conditions — Colitis, Ulcerative; Diabetes Mellitus, Insulin-Dependent, 12; Inflammatory Bowel Diseases | interventions — Hydroxychloroquine; Mesalamine

STUDY DESIGN:
Intervention Model Description: This is an Open Label study with blinded scorer for endoscopy and pathology reports.
Masking Description: The gastroenterologist who will review pre- and post-intervention endoscopy and pathology reports will be masked to any and all information about the study participants including disease severity and medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mesalamine and Hydroxychloroquine (Experimental): All participants will be on Mesalamine and Hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine; Drug: Mesalamine

INTERVENTIONS:
Drug: Hydroxychloroquine — 400mg of hydroxychloroquine per oral daily
Drug: Mesalamine — the participant will maintain their current standard of care dose which can range from 1.5g to 4.8g of mesalamine per oral daily

SUMMARY:
The objective of this study is to assess the efficacy of hydroxychloroquine (HCQ) when combined with Mesalamine in reducing clinical and histologic disease activity in patients who have active mild to severe Ulcerative Colitis (UC) and also to assess the immunological effects of hydroxychloroquine in this population. These outcomes will be evaluated both clinically and experimentally. In vitro, flow cytometry will be employed to measure the expression of CTLA-4 on activated CD4+CD25+CD127- Tregs from patients prior to treatment with HCQ, and then at the end of a 4 month follow up period. Suppression assays will be used to determine the functional capacity of the patient derived Tregs. Clinically, patients will be monitored for remission as defined by reduction in patient reported stool frequency and rectal bleeding (mayo sub-score 0 or 1) and endoscopically, by improvement in mucosal appearance (mayo sub-score 0 or 1), all objective measures in the mayo score.

DETAILED DESCRIPTION:
This is a single arm study to evaluate the efficacy and immunological effect of administering Hydroxychloroquine to patients of non-European ancestry who have active mild to severe Ulcerative Colitis in spite of Mesalamine therapy. 10 Participants will be recruited in Icahn School of Medicine at Mount Sinai and 10 in Emory University (20 across all sites).

Participants 18 years and above who identify as an individual of non-European ancestry with a diagnosis of Ulcerative Colitis will be approached for the study. Participants will be recruited from Mount Sinai IBD center prior to their standard of care endoscopy. Participants who meet the study's inclusion criteria i.e. If they currently have active disease, they will be able to receive the research medication.

Participants will be administered 400mg hydroxychloroquine tablets orally for four months in addition to Mesalamine. Pre and post medication clinical, endoscopic and immunological assessments will be compared. Participants will also be followed up with bi-monthly phone calls. Participants will have a post medication colonoscopy at the end of the 4 month period.

There is a risk of retinopathy and cardiomyopathy associated with long term use of the study drug at doses greater than 6.5mg/kg for more than 5 years. Participants will be screened for existing eye and heart disease and monitored pre and post medication for any new adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to severe active Ulcerative Colitis (confirmed by endoscopy at screening),
* Currently taking mesalamine,
* Be an individual of non-European ancestry.
* Adult 18 years and older

Exclusion Criteria

* Current use of biologics, steroids or other UC medications not including mesalamine.
* Presence of hepatic or renal insufficiency
* Pregnancy or lactation
* Known allergic reactions to components of the Hydroxychloroquine, Chloroquine or quinine products.
* Any pre-existing macular disease or cardiac disease.
* Treatment with another investigational drug or other intervention within 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in surface CTLA4 expression | baseline and 4 months
  Flow cytometry will be used to measure the expression of CTLA-4 on activated CD4+CD25+CD127- Tregs from patients prior to treatment with Hydroxychloroquine, and then at the end of a 4 month follow up period.

SECONDARY OUTCOMES:
Change in Endoscopy Mayo Score | baseline and 4 months
  Endoscopic remission will be measured using the mayo score which ranges from 0-3 with 0 meaning remission and 3 indication severe disease. Premedication endoscopy mayo score will be compared to end of study mayo score (at 4 months)
Change in Partial Mayo Score | baseline and 4 months
  Change in patient reported symptoms for stool frequency and rectal bleeding are objective measures in the partial mayo score which ranges from 0-3 for both parameters. A score of zero indicates remission and a score on 3 indicates severe disease. Pre-medication partial mayo scores will be compared to end of study partial mayo scores (at 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Judy H Cho, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Subra Kugathasan, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - Icahn School of Medicine at Mount Sinai/Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. To achieve aims in the approved proposal. Investigators should contact study team.